CLINICAL TRIAL: NCT07370701
Title: Evaluation of Passivity of Co-Cr Complete Arch Screw Retained Maxillary Prostheses Using Different Intraoral Scanners With the Aid of Auxiliary Geometric Device
Brief Title: Passivity of Full-Arch Co-Cr Maxillary Prostheses Using IOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Hamdy Abdel-Hay Dawood, Assistant Lecturer of Oral and Maxillofacial Prosthodontics, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: FDASU-RecID022318
Record Dates: First submitted 2026-01-13; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Passivity of Co-Cr Full-arch Maxillary Prostheses Via IOS
Keywords: intraoral scanner; Auxiliary geometric device; All on 4 maxilla; modified screw test

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open tray impression digitized by extraoral scanner (EO Group) (Experimental): A reference model was formed to check the accuracy of these 3 data acquisitions. The framework was designed and printed for the 3 groups to be placed in the reference model to check the passivity. Passivity was tested through modified 1-screw test by measuring the marginal gap by using a digital camera (add magnification). Each framework was placed in the patient's mouth to re-check the passivity, the best one was delivered to the patient after 4 months after osteointegration of the implants.
  Interventions: Other: Open tray impression technique
- Intraoral scan by using Medit i600 with AGD (M600 Group) (Experimental): A reference model was formed to check the accuracy of these 3 data acquisitions. The framework was designed and printed for the 3 groups to be placed in the reference model to check the passivity. Passivity was tested through modified 1-screw test by measuring the marginal gap by using a digital camera (add magnification). Each framework was placed in the patient's mouth to re-check the passivity, the best one was delivered to the patient after 4 months after osteointegration of the implants.
  Interventions: Other: Auxiliary Geometric Device (M600)
- Intraoral scan (CEREC Primescan; Dentsply Sirona) with AGD (PS Group) (Experimental): A reference model was formed to check the accuracy of these 3 data acquisitions. The framework was designed and printed for the 3 groups to be placed in the reference model to check the passivity. Passivity was tested through modified 1-screw test by measuring the marginal gap by using a digital camera (add magnification). Each framework was placed in the patient's mouth to re-check the passivity, the best one was delivered to the patient after 4 months after osteointegration of the implants.
  Interventions: Other: Auxiliary Geometric Device (PS)

INTERVENTIONS:
Other: Open tray impression technique — dental implant then open tray impression technique
  Arms: Open tray impression digitized by extraoral scanner (EO Group)
Other: Auxiliary Geometric Device (M600) — analyze the accuracy and passivity of complete-arch digital scans of completely edentulous arches by placing auxiliary geometric device
  Arms: Intraoral scan by using Medit i600 with AGD (M600 Group)
Other: Auxiliary Geometric Device (PS) — analyze the accuracy and passivity of complete-arch digital scans of completely edentulous arches by placing auxiliary geometric device
  Arms: Intraoral scan (CEREC Primescan; Dentsply Sirona) with AGD (PS Group)

SUMMARY:
Statement of the problem: Accurate digital scans of edentulous patients is challenging due to the absence of anatomic landmarks and geometric variations along the dental arch. Whether adding an auxiliary geometric device (AGD) will improve scanning is unclear.

Purpose: The aim of the study is to analyze the accuracy of complete-arch digital scans of completely edentulous arches by placing auxiliary geometric device.

Material and Methods: This in vivo study included patients who received complete arch screw-retained prostheses supported by 4 implants. Seven patients were randomly chosen; a dual scan protocol was performed for digital implant planning. Surgical guide and AGD were 3d printed. Three different data acquisition methods for each individual: Open tray impression digitized by extraoral scanner (EO Group), Intraoral scan by using Medit i600 with AGD (M600 Group), and Intraoral scan (CEREC Primescan; Dentsply Sirona) with AGD (PS Group). A reference model was formed to check the accuracy of these 3 data acquisitions. The framework was designed and printed for the 3 groups to be placed in the reference model to check the passivity. Passivity was tested through modified 1-screw test by measuring the marginal gap by using a digital camera (add magnification). Each framework was placed in the patient's mouth to re-check the passivity, the best one was delivered to the patient after 4 months after osteointegration of the implants.

ELIGIBILITY:
Inclusion Criteria:

* For a maxillary edentulous patient, the last extraction should be at least six months
* Non-smokers
* 50-70 years of age
* Have good oral hygiene and motivation.

Exclusion Criteria:

* Patients with major systemic diseases that may affect osseointegration
* Uncontrolled diabetes mellitus
* The need for extensive bone grafting in the planned implant site
* Pregnant female patient
* Under bisphosphonate treatment
* Limited mouth-opening for executing the guided implant surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
estimate the marginal gap using digital camera | after 4 months after osteointegration of the implants
  modified single screw test to check the passivity of the 3 frameworks in both the models and in the patient's mouth by radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin H Abd El Hay Dawoud, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Organization of African Unity Street,, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.prosdent.2018.09.017